CLINICAL TRIAL: NCT03811587
Title: Clinical Feasibility and Efficacy of Intermittent Use of a Fasting Mimicking Diet in the Treatment of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other); Health Holland (Other); IFOM ETS - The AIRC Institute of Molecular Oncology (Other); L-Nutra (Unknown)
Responsible Party: Principal Investigator, Hanno Pijl, Clinical Professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL63892.058.18 - P18.049
Record Dates: First submitted 2019-01-13; First posted 2019-01-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diet; Fasting
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fasting

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to the intervention or control group.
Masking Description: Only measurements by assessors will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Diabetes type 2 patients will take a fasting mimicking diet of 5 consecutive days a month, for a duration of 12 months. Besides this, they will receive usual diabetes care from the general practitioner.
  Interventions: Other: Fasting Mimicking diet
- Control group (No Intervention): Diabetes type 2 Patients will have no intervention, they will receive usual diabetes care from the general practitioner.

INTERVENTIONS:
Other: Fasting Mimicking diet — The fasting mimicking diet is though to activate the metabolism as fasting would do, although the diet does include several meals a day and more calories than conventional fasting diets.
  Arms: Treatment group

SUMMARY:
In this randomized, controlled, assessor blinded and prospective intervention study the investigators will evaluate the clinical feasibility and effectiveness of intermittent use of a fasting mimicking diet in patients with type 2 diabetes mellitus compared to usual care.

DETAILED DESCRIPTION:
100 individuals (men or women, ethnicity not specified) with type 2 diabetes and a BMI≥ 27, who are treated with diet only and have a HbA1c > 48, or who are treated with diet and a dose of metformin can participate in the study. Participants will use a fasting-mimicking diet for 5 consecutive days per month. For the other days, there are no regulations. During follow-up of one year, several study parameters will be measured including HbA1c and antidiabetic medication dosage.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Age > 17 years and <75 years
* Treatment with diet only and have a HbA1c > 48, or treatment with diet and metformin
* BMI ≥ 27

Exclusion Criteria:

* Recent myocardial infarction (< 6 months)
* Creatinine clearance < 30 ml/min/1,73m2 (MDRD)
* Pregnancy
* Contraindications for MRI
* Allergy for nuts, sesame, soya or another ingredient of the diet
* History of syncope with calorie restriction in the past
* Any significant other disease (at the discretion of the investigator)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Concentration of HbA1c | 12 months
Dosage of antidiabetic medication used | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanno Pijl, MD, PhD, Principal Investigator — Leiden Univerity Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

REFERENCES:
- [Derived] Schoonakker MP, van den Burg EL, van Peet PG, le Cessie S, Penny E, Numans ME, Pijl H, Lamb HJ. A fasting-mimicking diet programme reduces abdominal adipose tissue while preserving abdominal muscle mass in persons with type 2 diabetes. Nutr Metab Cardiovasc Dis. 2025 Oct;35(10):104111. doi: 10.1016/j.numecd.2025.104111. Epub 2025 Apr 30. PMID 40425403
- [Derived] van den Burg EL, Schoonakker MP, van Peet PG, le Cessie S, Numans ME, Pijl H, Lamb HJ. A fasting-mimicking diet programme reduces liver fat and liver inflammation/fibrosis measured by magnetic resonance imaging in patients with type 2 diabetes. Clin Nutr. 2025 Apr;47:136-145. doi: 10.1016/j.clnu.2025.02.017. Epub 2025 Feb 18. PMID 40020647
- [Derived] Roos PR, van den Burg EL, Schoonakker MP, van Peet PG, Numans ME, Pijl H, Westenberg JJM, Lamb HJ. Fasting-mimicking diet in type 2 diabetes reduces myocardial triglyceride content: A 12-month randomised controlled trial. Nutr Metab Cardiovasc Dis. 2025 Jul;35(7):103860. doi: 10.1016/j.numecd.2025.103860. Epub 2025 Jan 9. PMID 39934050
- [Derived] van den Burg EL, Schoonakker MP, Korpershoek B, Sommeling LE, Sturm CA, Lamb HJ, Pijl H, Numans ME, Adriaanse MA, van Peet PG. Self-initiated lifestyle changes during a fasting-mimicking diet programme in patients with type 2 diabetes: a mixed-methods study. BMC Prim Care. 2024 May 2;25(1):148. doi: 10.1186/s12875-024-02405-5. PMID 38698355
- [Derived] van den Burg EL, Schoonakker MP, van Peet PG, van den Akker-van Marle EM, Lamb HJ, Longo VD, Numans ME, Pijl H. Integration of a fasting-mimicking diet programme in primary care for type 2 diabetes reduces the need for medication and improves glycaemic control: a 12-month randomised controlled trial. Diabetologia. 2024 Jul;67(7):1245-1259. doi: 10.1007/s00125-024-06137-0. Epub 2024 Mar 28. PMID 38546821
- [Derived] van den Burg EL, Schoonakker MP, van Peet PG, van den Akker-van Marle ME, Willems van Dijk K, Longo VD, Lamb HJ, Numans ME, Pijl H. Fasting in diabetes treatment (FIT) trial: study protocol for a randomised, controlled, assessor-blinded intervention trial on the effects of intermittent use of a fasting-mimicking diet in patients with type 2 diabetes. BMC Endocr Disord. 2020 Jun 24;20(1):94. doi: 10.1186/s12902-020-00576-7. PMID 32580710